CLINICAL TRIAL: NCT02426762
Title: Use of a Quick Skin Sealant in Prevention of Surgical Site Infection After Laparoscopic Tumor Resection
Brief Title: Quick Skin Sealant in Closure of Surgical Wound After Laparoscopic Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wu Song, Director of Center of Gastrointestinal Surgery, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015[122]
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Complications of Surgical Procedures; Surgical Site Infection; Gastric Cancer; Colorectal Cancer; Gastrointestinal Stromal Tumor; Inflammatory Bowel Disease; Diverticula
Keywords: skin sealant; laparoscopic surgery; surgical site infection; wound healing
MeSH Terms: conditions — Surgical Wound Infection; Stomach Neoplasms; Colorectal Neoplasms; Gastrointestinal Stromal Tumors; Inflammatory Bowel Diseases; Diverticulum | interventions — Laparoscopy; Surgical Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sealant skin closure (Experimental): A quick skin sealant would be applied after laparoscopic surgery. All abdominal wounds are sealed by smearing the quick sealant (skin adhesive) twice. No additional gauges should be appended on wound areas. No further wound care should be applied unless any effusion or bleeding emerged around it.
  Interventions: Procedure: Laparoscopic surgery; Device: Skin sealant

INTERVENTIONS:
Procedure: Laparoscopic surgery — Various laparoscopic operations are performed for participants. Once all surgical procedures are successfully applied, surgical wounds which are associated with laparoscopic surgery would be sealed by a quick sealant. In all, the following surgical wounds would be left:
  * 4-5 trocar-produced incisions (5/10mm, minor incision)
  * 1 sample-retrieval incision (4-5cm, small incision)
Device: Skin sealant — After surgery, a quick skin sealant is applied in two layers of each wound to achieve skin closure. The sealant would be smeared twice on the wound area with 30 seconds of dry time required to form a firm seal.
  Other Names: Skin adhesive

SUMMARY:
The purpose of this study is to evaluate the short-term effect of sealant-assisted skin closure in prevention of surgical site infection after laparoscopic surgery.

DETAILED DESCRIPTION:
* Study design: A prospective cohort study
* Populations: Patients who have confirmed diagnosis of gastric cancer, colorectal cancer, gastrointestinal stromal tumor (GIST), inflammatory bowel disease and diverticula decide to receive laparoscopic surgery.
* Surgical techniques: laparoscopic operations should be successfully performed with a 3-4 cm minimal incision left for sample retrieval. In all, about five trocar-associated mini incisions and a sample-retrieval incision would be left prior to skin closure.
* Skin closure: A quick skin sealant would be applied to achieve a seal, without any suture made under the skin.
* Postoperative treatment: An enhanced recovery after surgery (ERAS) bundles would be applied for enrolled subjects. As for wound management, additional wound cares are not required. Patients can take shower at postoperative day 3 (POD3).
* Primary endpoint: The primary study endpoint is freedom from surgical site infection (SSI) within 30 days. The incidence of surgical site infection with the first 30 days after surgery would be explored.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent has been obtained from the patient.
* With confirmed diagnosis of gastric cancer, colorectal cancer, gastrointestinal stromal tumor, inflammatory bowel disease and diverticula.
* Endurable laparoscopic surgery without conversion.
* With moderate/good ECOG health rating (PS): 0-1 score.

Exclusion Criteria:

* Pregnant woman or lactating woman.
* With confirmed distant metastasis in liver, lung, bones, or other organs.
* Intolerable laparoscopic operation or converted to open surgery.
* With severe comorbidities, such as cardiovascular disease, chronic obstructive pulmonary disease, diabetes mellitus, and chronic renal dysfunction.
* With bad compliance or contraindication to enrollment.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
freedom from surgical site infection | within the first 30 days after laparoscopic surgery
  The study endpoint should be freedom from superficial surgical site infection (SSI) or deep SSI as defined by the Centers of Disease Control and Prevention National Nosocomial Infection Surveillance criteria.

SECONDARY OUTCOMES:
Length of hospital stay | an expected average of 4 weeks
  All participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Pain Scores on the Visual Analog Scale | within the first 30 days after laparoscopic surgery
  Postoperative pain would be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Song, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China